CLINICAL TRIAL: NCT01480245
Title: An Open-label Extension Study of the Long-term Safety, Tolerability and Efficacy of GSK2402968 in Subjects With Duchenne Muscular Dystrophy
Brief Title: Open Label Study of GSK2402968 in Subjects With Duchenne Muscular Dystrophy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was formally terminated given that GSK is not submitting an application for regulatory approval for drisapersen in Duchenne Muscular Dystrophy.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114349
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Muscular Dystrophies
Keywords: 968; Duchenne; DMD; drisapersen
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Continuous Dosing (Experimental): GSK2402968 6mg/kg/week
  Interventions: Drug: GSK2402968
- Intermittent Dosing (Experimental): GSK2402968 6mg/kg/week
  Interventions: Drug: GSK2402968
- Natural History Observation (No Intervention): The objective of this arm will be to explore DMD disease progression in a naturalistic setting once discontinuing active treatment

INTERVENTIONS:
Drug: GSK2402968 — 6mg/kg/week
  Arms: Continuous Dosing; Intermittent Dosing

SUMMARY:
The purpose of this study is to explore long-term safety, tolerability and efficacy of GSK2402968 in DMD subjects who previously participated in either DMD114117 or DMD114044.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in either DMD114117 or DMD114044
* Continued use of glucocorticoids
* Willing and able to comply with all protocol requirements
* Able to give informed consent
* French subjects: Eligible for inclusion only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Subject experienced a serious adverse event or who met safety stopping criteria that remains unresolved from DMD114117 or DMD114044, which in opinion of the investigator could have been attributable to study medication and is ongoing,
* Use of anticoagulants, antithrombotics or antiplatelet agents, previous treatment with investigational drugs,except GSK2402968, within 1 month of the first administration of study medication,
* Current or anticipated participation in any investigational clinical studies,
* History of significant medical disorder which may confound the interpretation of either efficacy or safety data e.g. current history of renal or liver disease/impairment, history of inflammatory disease.

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2011-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Differences between the 6MWD at baseline and Week 104 | 104 weeks

SECONDARY OUTCOMES:
Timed Function tests | 104 weeks
Muscle strength | 104 weeks
North Star Ambulatory Assessment Scores | 104 weeks
Creatine kinase Serum concentrations | 104 weeks
Pulmonary Function | 104 weeks
Pediatric Quality of Life Neuromuscular module | 104weeks
Clinician Global Impression of Improvement | 104 weeks
Health Utilities Index | 104 weeks
Frequency of accidental falls during 6 Minute Walk Distance test | 104 weeks
Functional Outcomes Assessment | 104 weeks
Time to major disease milestones | 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (57):
- GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires, Argentina
- Australia (2):
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Parkville, Victoria
- Belgium (2):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
- Brazil (6):
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Rio de Janeiro, Rio de Janeiro
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Ribeirão Preto, São Paulo
  - GSK Investigational Site, Santo André, São Paulo
  - GSK Investigational Site, São Paulo, São Paulo
- GSK Investigational Site, Sofia, Bulgaria
- Canada (3):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Chile (3):
  - GSK Investigational Site, Temuco, Región de La Araucania
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- Czechia (2):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Prague
- GSK Investigational Site, Koebenhavn Oe, Denmark
- France (8):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pau
  - GSK Investigational Site, Toulouse
- Germany (5):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Kiel, Schleswig-Holstein
- GSK Investigational Site, Budapest, Hungary
- GSK Investigational Site, Jerusalem, Israel
- Italy (4):
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Messina, Sicily
- Japan (4):
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
- Netherlands (2):
  - GSK Investigational Site, Leiden
  - GSK Investigational Site, Nijmegen
- GSK Investigational Site, Oslo, Norway
- GSK Investigational Site, Warsaw, Poland
- GSK Investigational Site, Moscow, Russia
- GSK Investigational Site, Seoul, South Korea
- Spain (3):
  - GSK Investigational Site, Esplugues de Llobregat. Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Valencia
- GSK Investigational Site, Kaohsiung City, Taiwan
- GSK Investigational Site, Ankara, Turkey (Türkiye)
- United Kingdom (2):
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne